CLINICAL TRIAL: NCT06322030
Title: Enhancing Mobility and Psychosocial Function in Obese Veterans Following Stroke Via Weight Loss and ExeRcise (EMPOWER)
Brief Title: Weight Loss and ExeRcise
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N4281-R; RX004281 (Other Grant/Funding Number: VA ORD RR&D); PRO0120848 (Other: IRB Approval)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: obesity; weight loss; quality of life
MeSH Terms: conditions — Stroke; Obesity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: The investigators will utilize a 2x2 factorial design to assess for changes in our outcomes over time between treatment groups.
Who Masked: Outcomes Assessor
Masking Description: The coordinator will not see group assignment, only a patient number which is entered into a software package.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diet (Experimental): 15 week weight management program
  Interventions: Dietary Supplement: FOCUS-15 Lifestyle Management Program
- Control (No Intervention): waitlist control
- Exercise (Experimental): exercise training
  Interventions: Behavioral: Exercise Training
- Diet + Exercise (Experimental): 15 week weight management program + exercise training
  Interventions: Dietary Supplement: FOCUS-15 Lifestyle Management Program; Behavioral: Exercise Training

INTERVENTIONS:
Dietary Supplement: FOCUS-15 Lifestyle Management Program — 15 week weight management program
  Other Names: Diet
  Arms: Diet; Diet + Exercise
Behavioral: Exercise Training — 15 weeks of progressive exercise training
  Arms: Diet + Exercise; Exercise

SUMMARY:
Weight loss interventions for neurologically health individuals have established benefits for improving physical and psychosocial function. The investigators believe that Veterans who have had a stroke would realize similar benefits and that the effects would be enhanced with concurrent exercise training. The investigators will study the effects of a 15-week lifestyle management program to determine if it can effectively improve some of the physical and psychosocial problems common in Veterans who have had a stroke.

DETAILED DESCRIPTION:
More than 2 million stroke survivors currently living in the U.S. are obese. Obesity is known to exacerbate age-related declines in function in these individuals and is associated with poorer clinical outcomes and quality of life. Weight-loss interventions are well-studied in neurologically healthy individuals and are shown to be effective for attenuating functional decline and improving quality of life. Despite these established benefits, there is currently an absence of studies investigating the effects of intentional weight loss on physical and/or psychosocial function in individuals following stroke. The investigators propose a trial aimed at Enhancing Mobility and Psychosocial function in Obese Veterans following stroke via Weight loss and ExeRcise (EMPOWER). This trial leverages a 15-week multidisciplinary approach to weight loss, via an existing lifestyle and weight management program, including caloric restriction, with or without concurrent supervised exercise training, as the catalyst by which remediation of physical and psychosocial impairments promote enhanced recovery in obese Veteran survivors of stroke. The investigators posit that successful weight loss will result in improvements in physical and psychosocial function (compared to control subjects) and that concurrent exercise will result in improved outcomes when compared to weight loss alone. The VHA 2010 Management of Stroke Rehabilitation Guidelines recommends that patients receive a formal rehabilitation assessment, the results of which should be used to determine the appropriate level of care and develop evidence-based interventions. However, without information regarding the effects of obesity and weight management on physical and psychosocial function as well as data on the long-term benefits of the program, evidence to guide decisions regarding the most appropriate approach to post-stroke rehabilitation for obese Veteran stroke survivors will remain elusive and recommendations for best available treatment cannot be met. Data from the proposed trial will have important clinical significance by determining the extent to which this type of program improves (or not) physical and psychosocial outcomes in Veterans following stroke and will provide a foundation for future studies aimed at establishing effectiveness of this approach to post-stroke care for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stroke at least 6 months prior
* BMI > 30 kg/m2
* Residual paresis in the lower extremity (Fugl-Meyer LE motor score <34)
* Ability to follow instructions, complete training and testing and to communicate exertion, pain and distress
* Provision of informed consent

  * Individuals who meet inclusion criteria must complete an exercise tolerance test and be cleared for participation by the study cardiologist

Exclusion Criteria:

* Unable to ambulate at least 150 feet or experienced intermittent claudication while walking
* Unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's
* Dementia
* Life expectancy <1 yr
* History of DVT or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest
* Current enrollment in a rehabilitation trial to enhance motor or psychosocial recovery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in distance walk in 6 minute Walk Test | approximately 15 weeks
  Distance walk in 6 minutes

SECONDARY OUTCOMES:
Change in daily step activity | approximately 15 weeks
  Steps per day
Change in score of Stroke Impact Scale (SIS) | approximately 15 weeks
  The 59 item SIS assesses post-stroke recovery in four psychosocial domains: social participation, emotion, communication, memory & thinking; two motor domains: mobility & strength, and overall activities of daily living as well as subjective extent of total recovery. Scores range from zero to 59, higher scores indicates better recovery.
Change in score of Sheehan Disability Scale (SDS) | approximately 15 weeks
  The SDS is a brief, 3-item patient rated assessment of the degree of disability/impairment in work/school, social life, and family life/home responsibilities. Scores on the SDS range from zero (unimpaired) to 30 (highly impaired).
Change in score of Inventory of Psychosocial Functioning (IPF) | approximately 15 weeks
  The IPF is an 80-item measure that more comprehensively indexes the domains assessed with the SDS but more finely resolves impairment. Each domain is scored from zero to 100 whither higher scores indicating higher impairment.

OTHER OUTCOMES:
Change in blood lipid profile | approximately 15 weeks
  The investigators will measure fasting glucose, triglycerides, and cholesterol (total, LDL and HDL)
Change in body composition in Dual-energy x-ray absorptiometry | approximately 15 weeks
  Body composition

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Gregory, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No